CLINICAL TRIAL: NCT00770224
Title: A Phase II Study of Iodine-131-Labeled Tositumomab in Combination With Cyclophosphamide, Doxorubicin, Vincristine, Prednisone and Rituximab Therapy for Patients With Advanced Stage Follicular Non-Hodgkin's Lymphoma
Brief Title: S0801 Iodine I 131 Tositumomab, Rituximab, and Combination Chemotherapy in Previously Untreated Stage II, Stage III, or Stage IV Follicular Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000615104; S0801 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; tositumomab I-131; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R-CHOP, tositumomab and rituximab (Experimental): Cyclophosphamide 750 mg/m2 IV Day 1 Doxorubicin 50 mg/m2 IV Day 1 Vincristine 1.4 mg/m2 IV Day 1 Prednisone 100 mg PO Days 1-5 Rituximab 375 mg/m2 IV Day 1 Q 21 Days x 6 Cycles
  Patients are restaged by CT scan. Unlabeled tositumomab antibody 450 mg IV within 12 after Cycle 6 of CHOP. Dosimetric dose 35 mg IV after infusion of unlabeled tositumomab antibody. Unlabeled tositumomab antibody 450 mg IV 7-14 days after dosimetric dose. Therapeutic dose 35 mg IV after infusion of unlabeled tositumomab antibody.
  Rituximab 375 mg/m2 IV q 3 months x 4 years beginning 1 year after registration.
  Interventions: Biological: rituximab; Biological: tositumomab; Drug: cyclophosphamide; Drug: doxorubicin; Drug: prednisone; Drug: vincristine; Radiation: tositumomab

INTERVENTIONS:
Biological: rituximab
Biological: tositumomab
Drug: cyclophosphamide
Drug: doxorubicin
Drug: prednisone
Drug: vincristine
Radiation: tositumomab
  Other Names: iodine I 131 tositumomab

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies, such as iodine I 131 tositumomab, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving a radiolabeled monoclonal antibody together with rituximab and combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects of giving iodine I 131 tositumomab together with rituximab and combination chemotherapy and to see how well it works in treating patients with previously untreated stage II, stage III, or stage IV follicular non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the response rate in patients with previously untreated stage II-IV follicular non-Hodgkin lymphoma treated with rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone (R-CHOP) in combination with iodine I 131 tositumomab.
* To evaluate the toxicity of this regimen in these patients.
* To estimate the 3-year progression-free survival rate in patients treated with this regimen.
* To estimate the 5-year progression-free and overall survival rate in patients treated with this regimen.
* To assess the safety profile of this regimen in these patients.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive R-CHOP* comprising rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with at least stable disease then proceed to consolidation therapy.

NOTE: *Patients receive R-CHOP in courses 1-4 and CHOP alone in courses 5 and 6.

* Consolidation therapy: Within 12 weeks after completion of induction therapy, patients receive tositumomab IV over 1 hour followed by a dosimetric dose of iodine I 131 tositumomab IV over 20 minutes. Patients then undergo whole body gamma camera scans over a 1-week period to determine the rate of total body clearance of radioactivity and the therapeutic dose of iodine I 131 tositumomab. Within 7-14 days after the dosimetric dose, patients receive tositumomab IV over 1 hour followed by a therapeutic dose of iodine I 131 tositumomab IV over 20 minutes. Patients with at least stable disease then proceed to maintenance therapy.
* Maintenance therapy: Beginning approximately 1 year after study entry and no more than 28 days after restaging, patients receive rituximab IV every 3 months for up to 4 years (16 courses) in the absence of disease progression or unacceptable toxicity.

After completion of maintenance therapy, patients are followed annually for up to 7 years. Patients who do not complete maintenance therapy are followed every 6 months for 2 years and then annually for up to 7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* grade 1, 2, or 3 follicular B-cell non-Hodgkin lymphoma meeting the following criteria:

  * Bulky stage II or stage III or IV disease
  * Diffuse large cell component must be < 25% of the biopsy
  * Confirmed cluster of differentiation antigen 20 (CD20) antigen-positive disease NOTE: *Needle aspiration or cytology are not considered adequate for pathology review
* Patient must have unilateral or bilateral bone marrow aspirate and biopsy performed within 42 days

  * Positive biopsy performed > 42 days but < 6 months allowed
* Previously untreated disease
* Bidimensionally measurable disease
* No clinical evidence of central nervous system (CNS) involvement by lymphoma

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Cardiac ejection fraction ≥ 45% by multigated acquisition scan (MUGA) or ECHO
* No significant cardiac abnormalities
* No known HIV positivity
* No requirement for continuous supplemental oxygen therapy
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer from which the patient is currently in complete remission
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 12 months after completion of maintenance therapy

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiotherapy, or antibody therapy for lymphoma
* No prior solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-04; Primary Completion 2017-04 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W. Friedberg, MD, Study Chair — James P. Wilmot Cancer Center; Oliver W. Press, MD, PhD, Study Chair — Fred Hutchinson Cancer Center; Lisa Rimsza, MD, Study Chair — University of Arizona
Locations (114):
- United States (114):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Falck Cancer Center at Arnot Ogden Medical Center, Elmira, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - U.T. Medical Center Cancer Institute, Knoxville, Tennessee
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Derived] Rutherford SC, Yin J, Pederson L, Perez Burbano G, LaPlant B, Shadman M, Li H, LeBlanc ML, Kenkre VP, Hong F, Blum KA, Dockter T, Martin P, Jung SH, Grant B, Rosenbaum C, Ujjani C, Barr PM, Unger JM, Cheson BD, Bartlett NL, Kahl B, Friedberg JW, Mandrekar SJ, Leonard JP. Relevance of Bone Marrow Biopsies for Response Assessment in US National Cancer Institute National Clinical Trials Network Follicular Lymphoma Clinical Trials. J Clin Oncol. 2023 Jan 10;41(2):336-342. doi: 10.1200/JCO.21.02301. Epub 2022 Jul 5. PMID 35787017
- [Derived] Barr PM, Li H, Burack WR, LeBlanc M, Smith SM, Gopal AK, Floyd JD, Persky DO, Press OW, Fisher RI, Friedberg JW. R-CHOP, radioimmunotherapy, and maintenance rituximab in untreated follicular lymphoma (SWOG S0801): a single-arm, phase 2, multicentre study. Lancet Haematol. 2018 Mar;5(3):e102-e108. doi: 10.1016/S2352-3026(18)30001-2. Epub 2018 Jan 26. PMID 29396094

RESULTS

PARTICIPANT FLOW:
Groups:
- R-CHOP+I-131 Tositumomab: Cyclophosphamide 750 mg/m2 IV Day 1 Doxorubicin 50 mg/m2 IV Day 1 Vincristine 1.4 mg/m2 IV Day 1 Prednisone 100 mg PO Days 1-5 Rituximab 375 mg/m2 IV Day 1 Q 21 Days x 6 Cycles
  Patients are restaged by CT scan. Unlabeled tositumomab antibody 450 mg IV within 12 after Cycle 6 of CHOP. Dosimetric dose 35 mg IV after infusion of unlabeled tositumomab antibody. Unlabeled tositumomab antibody 450 mg IV 7-14 days after dosimetric dose. Therapeutic dose 35 mg IV after infusion of unlabeled tositumomab antibody.
- Rituximab Maintenance: Rituximab 375 mg/m2 IV q 3 months x 4 years beginning 1 year after registration.
Period: Step 1: Induction
Arm/Group | R-CHOP+I-131 Tositumomab | Rituximab Maintenance
Started | 87 | 0
Eligible and Evaluable | 84 | 0
Completed | 73 | 0
Not Completed | 14 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Refusal unrelated to adverse event | 6 | 0
Not completed — Other reason not protocol specified | 2 | 0
Not completed — Ineligible | 2 | 0
Not completed — No protocol treatment given | 1 | 0
Period: Step 2: Maintenance
Arm/Group | R-CHOP+I-131 Tositumomab | Rituximab Maintenance
Started | 0 | 71
Eligible and Evaluable | 0 | 69
Completed | 0 | 41
Not Completed | 0 | 30
Not completed — Adverse Event | 0 | 10
Not completed — Refusal unrelated to adverse event | 0 | 8
Not completed — Progression/relapse | 0 | 1
Not completed — Death | 0 | 2
Not completed — Other reason not protocol specified | 0 | 7
Not completed — Ineligible | 0 | 2

BASELINE CHARACTERISTICS:
Population: Only eligible and evaluable patients were included in the analysis.
Arm/Group | R-CHOP+I-131 Tositumomab
Number analyzed (Participants) | 84
Age, Continuous [Median (Full Range); unit: years] | 52.3 [28.9 to 79.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 81
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 78
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 3-year Progression-free Survival (PFS)
Description: Measured from date of registration to date of first observation of progressive disease or death due to any cause. Progressive disease is ≥ 50% increase in the sum of products of greatest diameters (SPD) of target measurable nodal lesions over the smallest sum observed (over baseline if no decrease during therapy), or ≥ 50% increase in the greatest transverse diameter (GTD) of any node > 1 cm in shortest axis, or ≥ 50% increase in the SPD of other target measurable lesions (e.g., splenic or hepatic nodules) over the smallest sum observed. Appearance of any new bone marrow involvement; appearance of a new lesion/site; lymph nodes with the long axis is > 1.5 cm, or if the both the long and short axes are > 1 cm; in patients with no pretreatment PET scan or when the PET scan was positive before therapy, lesions should be PET positive; or death due to disease without prior documentation of progression.
Time Frame: 0-3 years
Population: Eligible and evaluable patients were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- R-CHOP+I-131 Tositumomab Followed by Rituximab Maintenance: Cyclophosphamide 750 mg/m2 IV Day 1 Doxorubicin 50 mg/m2 IV Day 1 Vincristine 1.4 mg/m2 IV Day 1 Prednisone 100 mg PO Days 1-5 Rituximab 375 mg/m2 IV Day 1 Q 21 Days x 6 Cycles
  Patients are restaged by CT scan. Unlabeled tositumomab antibody 450 mg IV within 12 after Cycle 6 of CHOP. Dosimetric dose 35 mg IV after infusion of unlabeled tositumomab antibody. Unlabeled tositumomab antibody 450 mg IV 7-14 days after dosimetric dose. Therapeutic dose 35 mg IV after infusion of unlabeled tositumomab antibody.
  Rituximab 375 mg/m2 IV q 3 months x 4 years beginning 1 year after registration.
Arm/Group | R-CHOP+I-131 Tositumomab Followed by Rituximab Maintenance
Number analyzed (Participants) | 84
percentage of participants | 90 [81.9 to 95.1]

2. Secondary Outcome: 5-year Progression-free Survival
Description: as for outcome 1
Time Frame: 0-5 years
Population: Eligible and evaluable patients were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-CHOP+I-131 Tositumomab Followed by Rituximab Maintenance
Number analyzed (Participants) | 84
percentage of participants | 85 [74.8 to 90.7]

3. Secondary Outcome: 5-year Overall Survival
Description: Measured from date of registration to date of death due to any cause. Patients last known to be alive and are censored at date of last contact.
Time Frame: 0-5 years
Population: Eligible and evaluable patients were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-CHOP+I-131 Tositumomab Followed by Rituximab Maintenance
Number analyzed (Participants) | 84
percentage of participants | 94 [86.3 to 97.5]

4. Secondary Outcome: Response Rate
Description: Complete (CR), complete unconfirmed (CRU) and partial responses (PR). CR is complete disappearance of all measurable and non-measurable disease with the exception of the following. Positron emission tomography (PET) must be negative if no pre-treatment PET scan or when the PET was positive before therapy. If the PET scan was negative before therapy, all nodal masses must have regressed. no new lesions; previously enlarged organs must have regressed in size; and if bone marrow positive at baseline, it must be negative. PR is ≥ 50% decrease in sum of products of greatest diameters (SPD) for up to six identified dominant lesions identified at baseline; no new lesions; no increase in the size of liver, spleen or other nodes; and splenic and hepatic nodules must have regressed in size by at least 50% in SPD. In patients with no pre-treatment PET scan or when the PET scan was positive before therapy, PET should be positive in at least one previously involved site.
Time Frame: up to 5 years (1 year induction + 4 years maintenance therapy) or time of disease progression
Population: Eligible and evaluable patients were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | R-CHOP+I-131 Tositumomab Followed by Rituximab Maintenance
Number analyzed (Participants) | 84
Participants
  Complete Response | 61
  Patital Response | 22
  Assessment Inadequate | 1

5. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: up to 5 years (1 year induction + 4 years maintenance therapy) or time of disease progression.
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 4.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | R-CHOP+I-131 Tositumomab | Rituximab Maintenance
Number analyzed (Participants) | 84 | 69
Participants
  Albumin, serum-low (hypoalbuminemia) | 1 | 0
  Allergic reaction/hypersensitivity | 2 | 0
  Anorexia | 1 | 0
  Cough | 1 | 1
  Diarrhea | 1 | 0
  Dyspnea (shortness of breath) | 1 | 0
  Enteritis (inflammation of the small bowel) | 0 | 1
  Fatigue (asthenia, lethargy, malaise) | 8 | 1
  Febrile neutropenia | 14 | 0
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 2 | 0
  Glucose, serum-high (hyperglycemia) | 4 | 0
  Hemoglobin | 6 | 0
  Hypotension | 2 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Bladder | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Catheter-rel | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Dental-tooth | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Lymphatic | 2 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Pharynx | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - UTI | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Upper airway | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Wound | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Mid ear | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Sinus | 0 | 1
  Left ventricular systolic dysfunction | 1 | 1
  Leukocytes (total WBC) | 34 | 0
  Lymphopenia | 25 | 4
  Mood alteration - anxiety | 0 | 1
  Mood alteration - depression | 0 | 1
  Muscle weakness, not d/t neuropathy - body/general | 1 | 1
  Nasal cavity/paranasal sinus reactions | 0 | 1
  Nausea | 3 | 0
  Neuropathy: motor | 1 | 0
  Neuropathy: sensory | 6 | 0
  Neutrophils/granulocytes (ANC/AGC) | 48 | 1
  Opportunistic inf associated w/gt=Gr 2 lymphopenia | 1 | 0
  Pain - Abdomen NOS | 1 | 0
  Pain - Bone | 1 | 0
  Pain - Head/headache | 1 | 0
  Pain - Muscle | 1 | 0
  Pain-Other (Specify) | 0 | 1
  Platelets | 17 | 0
  Pulmonary hypertension | 0 | 1
  Restrictive cardiomyopathy | 0 | 1
  Secondary Malignancy-poss rel to cancer Tx | 0 | 1
  Sodium, serum-low (hyponatremia) | 1 | 0
  Syncope (fainting) | 1 | 0
  Thrombosis/thrombus/embolism | 1 | 0
  Valvular heart disease | 0 | 1
  Vasovagal episode | 0 | 1
  Vision-blurred vision | 1 | 0
  Vomiting | 2 | 0
  Weight loss | 1 | 0

ADVERSE EVENTS:
Time Frame: up to 5 years (1 year induction + 4 years maintenance therapy) or time of disease progression.
Arm/Group | R-CHOP+I-131 Tositumomab | Rituximab Maintenance
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/84 | 1/69
Other Adverse Events (participants affected / at risk) | 84/84 | 66/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R-CHOP+I-131 Tositumomab (N=84) | Rituximab Maintenance (N=69)
Secondary Malignancy-poss rel to cancer Tx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | R-CHOP+I-131 Tositumomab (N=84) | Rituximab Maintenance (N=69)
Febrile neutropenia (Blood and lymphatic system disorders) | 15 | 0
Hemoglobin (Blood and lymphatic system disorders) | 56 | 18
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 4
Palpitations (Cardiac disorders) | 2 | 4
Thyroid function, high (Endocrine disorders) | 0 | 4
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 2 | 7
Vision-blurred vision (Eye disorders) | 6 | 4
Constipation (Gastrointestinal disorders) | 40 | 9
Diarrhea (Gastrointestinal disorders) | 18 | 15
Heartburn/dyspepsia (Gastrointestinal disorders) | 15 | 5
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 6 | 0
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 10 | 2
Nausea (Gastrointestinal disorders) | 58 | 16
Pain - Abdomen NOS (Gastrointestinal disorders) | 23 | 10
Vomiting (Gastrointestinal disorders) | 21 | 5
Edema: limb (General disorders) | 12 | 7
Fatigue (asthenia, lethargy, malaise) (General disorders) | 70 | 42
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 7 | 3
Pain-Other (General disorders) | 9 | 14
Rigors/chills (General disorders) | 15 | 2
Allergic reaction/hypersensitivity (Immune system disorders) | 14 | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Bronchus (Infections and infestations) | 0 | 4
Inf w/normal ANC or Gr 1-2 neutrophils - Sinus (Infections and infestations) | 0 | 12
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 3 | 5
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 7 | 4
Infection with unknown ANC - Sinus (Infections and infestations) | 0 | 9
Infection-Other (Infections and infestations) | 4 | 7
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 15 | 11
AST, SGOT (Investigations) | 14 | 10
Alkaline phosphatase (Investigations) | 9 | 5
Bilirubin (hyperbilirubinemia) (Investigations) | 4 | 8
Creatinine (Investigations) | 8 | 10
Leukocytes (total WBC) (Investigations) | 60 | 31
Lymphopenia (Investigations) | 36 | 32
Metabolic/Laboratory-Other (Investigations) | 10 | 10
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 56 | 9
Platelets (Investigations) | 58 | 26
Weight gain (Investigations) | 7 | 10
Weight loss (Investigations) | 8 | 9
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 14 | 5
Anorexia (Metabolism and nutrition disorders) | 25 | 8
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 12 | 6
Dehydration (Metabolism and nutrition disorders) | 6 | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 35 | 22
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 6 | 4
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 7 | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 5 | 4
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 12 | 7
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 13 | 5
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 5 | 1
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 10 | 3
Pain - Back (Musculoskeletal and connective tissue disorders) | 12 | 11
Pain - Bone (Musculoskeletal and connective tissue disorders) | 11 | 4
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 6 | 6
Pain - Joint (Musculoskeletal and connective tissue disorders) | 13 | 18
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 16 | 11
Dizziness (Nervous system disorders) | 15 | 8
Neuropathy: sensory (Nervous system disorders) | 48 | 15
Pain - Head/headache (Nervous system disorders) | 24 | 8
Taste alteration (dysgeusia) (Nervous system disorders) | 16 | 0
Insomnia (Psychiatric disorders) | 24 | 13
Mood alteration - anxiety (Psychiatric disorders) | 18 | 10
Mood alteration - depression (Psychiatric disorders) | 7 | 14
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 21
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 19 | 8
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 4 | 5
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 46 | 3
Nail changes (Skin and subcutaneous tissue disorders) | 5 | 3
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 8 | 5
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 5 | 2
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 13 | 10
Hot flashes/flushes (Vascular disorders) | 9 | 10
Hypertension (Vascular disorders) | 3 | 10
Hypotension (Vascular disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT00770224/Prot_SAP_ICF_000.pdf